CLINICAL TRIAL: NCT06748196
Title: Awareness Among Physiotherapists of Khyber Pakhtunkhwa About the Effectiveness of Sensory Integration Therapy on Cerebral Palsy Population.
Brief Title: Awareness Among Physiotherapists About Effectiveness of Sensory Integration Therapy on Cerebral Palsy Population.
Status: Recruiting | Type: Observational
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Other Study IDs: REC/RCR/AHS/24/0719
Record Dates: First submitted 2024-11-03; First posted 2024-12-27 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2025-01

CONDITIONS: Cerebral Palsy (CP)
Keywords: Cerebral Palsy; Sensory Integration Therapy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pediatric Physiotherapists: • Physical Therapists working across Khyber Pakhtunkhwa representative of all divisions of the province. • Physical Therapists working as clinicians or working in healthcare vicinities from at least 2 years.

SUMMARY:
The study is to interrogate the awareness level of physiotherapists that are working in the region of KHYBER PAKHTUNKHWA, to access whether they know about sensory integration therapy or they use it for the patients of cerebral palsy in their treatment plan or not.

DETAILED DESCRIPTION:
The study title is ''AWARENESS AMONG PHYSICAL THERAPISTS OF KHYBER PAKHTUNKHWA ABOUT THE EFFECTIVENESS OF SENSORY INTEGRATION THERAPY ON CEREBRAL PALSY POPULATION.' it is a cross-sectional study that will be conducted in the province of Khyber Pakhtunkhwa, Pakistan. The data will be conducted by 110 physical therapists on a self designed tool, that will allow us to know about the awareness among the physical therapist of this particular region to know if they are using sensory integration therapy in the treatment plan of the children suffering from cerebral palsy to know whether the sensory issues are being addressed over there by this therapy or not. Another purpose of this study is to make the therapists aware about sensory integration therapy and its efficacy in treating sensory processing and sensory integration issues present in the children that are suffering from cerebral palsy. The data will be collected by the physical therapists that are currently working in various hospitals of Khyber Pakhtunkhwa located in different regions of the province.

ELIGIBILITY:
Inclusion Criteria:

* Physical Therapists working across Khyber Pakhtunkhwa representative of all divisions of the province.
* Physical Therapists working as clinicians or working in healthcare vicinities from at least 2 years.

Exclusion Criteria:

* Non practicing Physical Therapists
* Freshly graduated Physical Therapists
* Physical Therapists working in areas other than Khyber Pakhtunkhwa

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Physical Therapists of Khyber Pakhtunkhwa
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-09-25 (Actual); Primary Completion 2025-01-05 (Estimated); Study Completion 2025-01-10 (Estimated)

PRIMARY OUTCOMES:
Survey tool awareness of Physical Therapists about sensory integration therapy | 60 minutes
  Survey was conducted through adapted questionnaire among the physical therapists of Khyber Pakhtunkhwa

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Shafique Akhtar, MS*, Principal Investigator — Riphah International Lahore
Locations (1):
- Riphah International University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Warutkar VB, Krishna Kovela R. Review of Sensory Integration Therapy for Children With Cerebral Palsy. Cureus. 2022 Oct 26;14(10):e30714. doi: 10.7759/cureus.30714. eCollection 2022 Oct. PMID 36439588